CLINICAL TRIAL: NCT05691491
Title: A Phase 1/2 Trial Evaluating the Combination of Temozolomide and the Ataxia Telangiectasia and Rad3-Related Inhibitor M1774
Brief Title: Testing the Combination of the Anti-Cancer Drugs Temozolomide and M1774 to Evaluate Their Safety and Effectiveness
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-10211; NCI-2022-10211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10572 (Other: Yale University Cancer Center LAO); 10572 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2023-01-18; First posted 2023-01-20 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Advanced Microsatellite Stable Colorectal Carcinoma; Hematopoietic and Lymphatic System Neoplasm; Metastatic Malignant Solid Neoplasm; Metastatic Microsatellite Stable Colorectal Carcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tuvusertib, temozolomide) (Experimental): Patients receive tuvusertib PO QD) on days 1-7 and temozolomide PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and MRI as well as collection of blood samples throughout the trial. Patients also undergo a biopsy at baseline and may undergo one on study and/or at time of progression.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Temozolomide; Drug: Tuvusertib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Temozolomide — Given orally (PO)
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Tuvusertib — Given PO
  Other Names: ATR Kinase Inhibitor M1774; M 1774; M-1774; M1774

SUMMARY:
This phase I/II trial studies the side effects and best dose of temozolomide and M1774 and how well they works in treating patients with cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and may have spread to nearby tissue, lymph nodes, or distant parts of the body (advanced). Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid (DNA) and may kill tumor cells and slow down or stop tumor growth. M1774 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Adding M1774 to temozolomide may shrink or stabilize cancer for longer than temozolomide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose of the combination of temozolomide (TMZ) and tuvusertib (M1774).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the overall response rate. III. To estimate progression free survival. IV. To estimate overall survival. V. To determine the recommended phase 2 dose of the combination of TMZ and M1774.

EXPLORATORY OBJECTIVES:

I. Correlate MGMT promoter hypermethylation, MGMT expression and tumor-infiltrating lymphocytes (TILs) with efficacy endpoints of response rate, progression free survival, and overall survival.

II. Assess pre and post treatment tumor biopsies for changes in tumor mutational burden, tumor associated neo-antigens and microsatellite status by whole exome sequencing.

III. Measure changes in peripheral blood mononuclear cell populations with treatment.

IV. Assess liquid biopsies by circulating tumor (ct)DNA for changes in tumor mutational burden and microsatellite status by whole exome sequencing.

OUTLINE: This is a phase I, dose-escalation study of temozolomide and tuvusertib followed by a phase II study.

Patients receive tuvusertib orally (PO) once daily (QD) on days 1-7 and temozolomide PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan and magnetic resonance imaging (MRI) as well as collection of blood samples throughout the trial. Patients also undergo a biopsy at baseline and may undergo one on study and/or time of progression.

After completion of study treatment, patients are followed up at 4 weeks, and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of metastatic advanced cancer.
* In dose escalation, any solid tumor patients with either O6-methylguanine DNA methyltransferase (MGMT) promoter hypermethylation positivity on testing / pre-screening of archival tissue OR an extracranial solid tumor where TMZ is considered a standard of care per National Comprehensive Cancer Network (NCCN) guidelines (neuroendocrine tumor, small cell lung cancer, melanoma or soft tissue sarcoma). The tumor lesion must be safely accessible to a mandatory biopsy. Patients with MGMT promoter hypermethylated colorectal cancer must be mismatch repair proficient / microsatellite stable.
* In phase 2, only patients with mismatch repair proficient / microsatellite stable colorectal cancer that have MGMT promoter hypermethylation positivity on pre-screening of archival tissue will be eligible.
* In dose escalation, patients must have progressed after treatment with all available therapies including immunotherapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment. Patients may not have previously received temozolomide or an ataxia telangiectasia and rad3-related (ATR) inhibitor.
* For patients with mismatch repair proficient / microsatellite stable colorectal cancer in the phase 2 portion, patients must have received prior therapy with 1 or more systemic therapies in the metastatic setting that includes 5-fluorouracil, irinotecan, and oxaliplatin. Patients with microsatellite stable colorectal cancer (mCRC) need to have had exposure, unless contraindicated, to all 3 of oxaliplatin, irinotecan, and fluoropyrimidine (FP).

The use of 5-fluorouracil and oxaliplatin in the adjuvant setting is acceptable, provided the development of metastatic disease was less than 6 months after the completion of adjuvant therapy.

Patients with a prior hypersensitivity reaction to oxaliplatin in the adjuvant setting do not require retreatment in the metastatic setting.

* Age >=18 years. Because no dosing or adverse event data are currently available on the use of M1774 in combination with temozolomide in patients < 18 years of age, children are excluded from this study.
* Measurable disease on CT and/or MRI per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (or Karnofsky >= 60%).
* Hemoglobin >=10 g/dL (No blood transfusions are allowed within 14 days of cycle 1 day 1 [C1D1]).
* White blood cells (WBC) > 3 x 10^9/L.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 100,000/mcL.
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine-aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 3 x institutional ULN except for when liver metastases are present, in which case they must be =< 5 x institutional ULN.
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for 4 weeks.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* The effects of M1774 on the developing human fetus are unknown. For this reason and because ATR inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 6 months after completion of M1774 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of M1774 administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and neuropathy, which may be =< grade 2.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to M1774 or temozolomide, including dacarbazine.
* Patients with uncontrolled intercurrent illness.
* Pregnant women are excluded from this study because M1774 is an ATR inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M1774 breastfeeding should be discontinued if the mother is treated with M1774. These potential risks also apply to temozolomide.
* Patients with a prior history of ataxia telangiectasia.
* Patients who are not able to swallow orally administered medication or have gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients who cannot discontinue proton-pump inhibitors (PPIs) while taking M1774. H-2 receptor antagonists are allowed but should not be taken within 12 hours before or 2 hours after M1774. Antacids are also allowed, but should not be taken 2 hours before 2 hours after M1774.
* Extensive RT involving greater than 30% of the bone marrow is not permitted during the study.
* A Fridericia's correction formula (QTcF) > 480 ms is exclusionary given the potential for QT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity and the maximum tolerated dose | Up to 28 days
  Defined as adverse events meeting the criteria that are at least "possibly related" to TMZ or M1774. Dose limiting toxicity for temozolomide in combination with M1774 and the maximum tolerated dose or maximum safe dose. Will consider ten dose levels (dose level -2, -1, 1, 2, 3, 4, 5, 6, 7, 8). The Bayesian Optimal Interval (BOIN) design based on the cumulative number of patients who experience a dose-limiting toxicity (DLT) at the current dose level will be used to guide dose escalation.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Will report the ORR and corresponding 2-sided 90% exact confidence intervals using the Clopper-Pearson method.
Progression free survival (PFS) | From start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
  Will be estimated using Kaplan-Meier method. Median survival times will be estimated. The confidence intervals for the median will be calculated. Log-rank test will be used to compare the PFS between the MGMT+ and MGMT- group.
Overall survival (OS) | Up to 2 years
  Will be estimated using Kaplan-Meier method. Median survival times will be estimated. The confidence intervals for the median will be calculated. Log rank test will be used to compare the OS between the MGMT+ and MGMT- group.
Rate of >= grade 3 adverse events (AE) | Up to 2 years
  The revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cecchini, Principal Investigator — Yale University Cancer Center LAO
Locations (23):
- United States (23):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm